CLINICAL TRIAL: NCT06383793
Title: Comparative Analysis of Short-Term Therapeutic Effects Between the π-Shaped and Overlap Methods for Esophagogastrostomy in Totally Laparoscopic Total Gastrectomy
Status: Recruiting | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Daorong Wang, Dr, Northern Jiangsu People's Hospital
Other Study IDs: Northjiangsu000
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — EXOSC10 protein, human

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- overlap
  Interventions: Procedure: overlap
- Π
  Interventions: Procedure: overlap

INTERVENTIONS:
Procedure: overlap — Π

SUMMARY:
As of now, although the safety of π-shaped anastomosis and the overlap method has been separately discussed in different contexts, there have been few studies considering a direct comparison of the results of these two methods.

This article aims to explore the differences in the short-term therapeutic effects, surgical effectiveness, and safety between laparoscopic total gastrectomy with esophagogastrostomy using the overlap method and the π-shaped method. The goal is to provide new reference points for surgeons in the clinical decision-making process regarding the choice of anastomotic techniques during totally laparoscopic total gastrectomy.

ELIGIBILITY:
Inclusion Criteria:(1) preoperative confirmation through electronic gastroscopy and enhanced CT that the lesion was situated in the fundus, middle and upper third of the gastric body, or the entire stomach; (2) postoperative pathology confirming adenocarcinoma; (3) utilization of either overlap esophagojejunal anastomosis or π-shaped anastomosis in total laparoscopic total gastrectomy.

-

Exclusion Criteria:(1) patients with severe preoperative cardiac, hepatic, renal, and pulmonary complications; (2) preoperative neoadjuvant chemotherapy; (3) a history of previous abdominal surgery; (4) patients requiring combined resection due to infiltration of other organs during the operation; (5) patients with incomplete pathological or clinical data. All patients signed informed consent.

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: preoperative confirmation through electronic gastroscopy and enhanced CT that the lesion was situated in the fundus, middle and upper third of the gastric body, or the entire stomach
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
1 year survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Yifan Cheng, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes